CLINICAL TRIAL: NCT00276835
Title: A Pilot Study of the Effect of Genistein in Combination With High-Dose Interleukin-2 on Cell Expansion and Gene Expression in Patients With Metastatic Melanoma or Renal Cell Carcinoma
Brief Title: Genistein and Interleukin-2 in Treating Patients With Metastatic Melanoma or Kidney Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Timothy Kuzel, Timothy Kuzel, MD, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 04V1; NU-04V1; CHIR-NU-04V1; NU-IRB-0310-083
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: recurrent renal cell cancer; clear cell renal cell carcinoma; stage IV renal cell cancer; recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — Interleukin-2; aldesleukin; Genistein; Isoflavones

ARMS (1):
- Genistein and Interleukin-2 (Experimental)
  Interventions: Biological: High-dose interleukin-2; Dietary Supplement: genistein

INTERVENTIONS:
Biological: High-dose interleukin-2 — Administered days 1-5, and 15-19; the patient will receive 600,000 IU/kg IL-2 by intravenous infusion over 15 minutes every 8 hours (on day 1 and day 15, patients will receive a maximum of 2 doses per day; on all other days in the cycle patients will receive a maximum of 3 doses per day)
  Other Names: IL-2; Aldesleukin; Proleukin
Dietary Supplement: genistein — Starting on day 10 and continuing through day 19, genistein will be administered orally at a dose of 600mg/day in two divided doses (i.e. 300mg po bid x 10 days)
  Other Names: isoflavone

SUMMARY:
RATIONALE: Genistein may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Interleukin-2 may stimulate the white blood cells, including natural killer cells, to kill melanoma or kidney cancer cells. Giving genistein together with interleukin-2 may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving genistein together with interleukin-2 works in treating patients with metastatic melanoma or kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Measure the differences in peak and duration of the expansion of circulating CD4-positive, CD8-positive, and CD4-, CD25-, and CD56-positive cells (dim and bright) at different time points during therapy with interleukin-2 (IL-2) alone and plus genistein in patients with metastatic malignant melanoma or renal clear cell carcinoma.

Secondary

* Evaluate the differences in peripheral blood mononuclear cell gene expression following high-dose IL-2 with and without genistein and compare to baseline.
* Determine the overall response rate (partial and complete) in patients treated with these regimens.
* Determine the safety and toxic effects of these regimens in these patients.
* Determine the time to progression in patients treated with these regimens.

OUTLINE: This is a pilot study.

Patients receive high-dose interleukin-2 IV over 15 minutes twice daily on days 1 and 15 and 3 times daily on days 2-5 and 16-19. Patients also receive oral genistein twice daily on days 10-19.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Documented histologically confirmed malignant melanoma or renal clear cell carcinoma

  * Metastatic disease
* At least 1 measurable lesion that can be accurately measured in at least one dimension with longest diameter > 20 mm using conventional techniques OR > 10 mm with spiral CT scan

  * If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology
  * Clinical lesions will only be considered measurable when they are superficial (e.g., skin nodules or palpable lymph nodes)
  * The following are considered non-measurable lesions:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Cystic lesions
    * Abdominal masses that are not confirmed and followed by imaging techniques
* No CNS metastases by CT scan or MRI

PATIENT CHARACTERISTICS:

* ECOG performance status < 2
* Life expectancy ≥ 4 months
* Serum creatinine < 2.0 mg/dL OR creatinine clearance > 50 mL/min
* Bilirubin normal
* Platelets > 100,000/mm³
* WBC > 3,500/mm³
* No evidence of congestive heart failure
* No symptom of coronary artery disease
* No serious cardiac arrhythmias
* A pretreatment cardiac stress test must be performed within 42 days of IL-2 treatment if any cardiac symptoms present (patients with documented ischemia on the pretreatment cardiac stress test will be excluded from the study)
* Adequate pulmonary reserve

  * FEV_1 > 75% of predicted
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test
* No known HIV-positive patients
* No evidence of active infection requiring antibiotic therapy
* No contraindication to treatment with pressor agents
* No significant medical disease which, in the opinion of the investigator, may interfere with completion of the study
* No history of another malignancy other than basal cell skin cancer within 5 years

PRIOR CONCURRENT THERAPY:

* Recovered from all toxic effects of prior therapy
* No radiotherapy, chemotherapy, or immunotherapy in the 4 weeks prior to the first dose of the study treatment
* No systemic corticosteroids in the 4 weeks prior to treatment
* No previous investigational agent within 4 weeks prior to the start of the study
* No prior interleukin-2 therapy
* No organ allografts allowed
* No concurrent radiotherapy, chemotherapy, or immunotherapy
* No concurrent corticosteroids
* No concurrent chronic medication for asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-11; Primary Completion 2007-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Differences in peak and duration of the expansion of circulating CD4+, CD8+, and CD4+, CD25+, and CD56+ cells (dim and bright) | Days 1, 8, 10, 15, 22, and 24 of treatment

SECONDARY OUTCOMES:
Circulating plasma levels of TGF-beta | Prior to and at end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States